CLINICAL TRIAL: NCT00505102
Title: Efficacy and Safety of Everolimus to SAve REnal Function (SAREFU) in Long Term Heart Transplanted Patients
Brief Title: Safe Renal Function In Long Term Heart Transplanted Patients
Acronym: SAREFU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Roberto Fiocchi, Ospedali Riuniti Bergamo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAREFU123
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Kidney Diseases; Heart Transplantation
Keywords: Kidney Diseases; Heart Transplantation; Everolimus; Cyclosporine Toxicity
MeSH Terms: conditions — Kidney Diseases | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — cyclosporine dose reduced of 50% after introduction of everolimus

SUMMARY:
The purpose of this study is to verify whether the reduction of cyclosporine dosages associated with Everolimus administration may improve renal function as compared to patients maintained on standard immunosuppressive therapy

ELIGIBILITY:
Inclusion Criteria:

* Heart Transplant patients with more than 1 year of follow-up
* Creatinine lower than 3.5 mg/dl
* GFR Higher than 20 ml/min (calculated with Cockcroft-Gault formula)
* Cyclosporine in maintenance immunosuppressive therapy
* Patient must be able to sign an approve informed consent
* Prior History of acute rejection within the last 3 months
* Females of childbearing age may be included if pregnancy is excluded and acceptable contraception measures are used

Exclusion Criteria:

* Patients who are recipients of multiple organ transplants
* Prior or current use of sirolimus or everolimus
* History of acute rejection within the last 6 months
* Coronary Artery Bypass Surgery or other cardiac surgery in the past 3 months
* Patient not able to attend all follow-up evaluations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Renal function Evaluated measuring Creatinine, Creatinine Clearance (MDRD and Cockcroft-Gault) and Urinary excretion of Protein, albumin and alpha-1-microglobulin | 2 years

SECONDARY OUTCOMES:
All cause mortality, infections, incidence of acute myocardial rejection, Heart Failure, Chronic Rejection, Mace | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fiocchi, MD PhD, Study Director — Heart Transplant Center Ospedali Riuniti Bergamo
Locations (2):
- Italy (2):
  - Heart Transplant Center Ospedali Riuniti, Bergamo
  - Heart Transplantad Center OspedaliRiuniti Bergamo, Bergamo

REFERENCES:
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Rothenburger M, Teerling E, Bruch C, Lehmkuhl H, Suwelack B, Bara C, Wichter T, Hinder F, Schmid C, Stypmann J. Calcineurin inhibitor-free immunosuppression using everolimus (Certican) in maintenance heart transplant recipients: 6 months' follow-up. J Heart Lung Transplant. 2007 Mar;26(3):250-7. doi: 10.1016/j.healun.2007.01.017. PMID 17346627